CLINICAL TRIAL: NCT02594553
Title: Optimizing Management and Medication of Febrile Children in Out-of-hours Primary Care: the CHILI Cluster Randomised Trial
Brief Title: Optimizing Management and Medication of Febrile Children in Out-of-hours Primary Care: CHILI Cluster RCT
Acronym: CHILI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZonMw GGG - 836021022
Record Dates: First submitted 2015-10-26; First posted 2015-11-03 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2015-10

CONDITIONS: Antibiotic Prescriptions; Infection
Keywords: Antibiotics; Children; General Practitioner; GP; After-hours care; Out-of-hours care; Booklet; Primary Health Care; Child
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): All GPs working at the participating GP out-of-hours centres that are in the intervention group will use the GP-parent information-exchange tool (interactive booklet).
  Interventions: Behavioral: GP-parent information-exchange tool
- Control (No Intervention): All GPs working at the participating GP out-of-hours centres that are in the control group will provide care as usual.

INTERVENTIONS:
Behavioral: GP-parent information-exchange tool — The booklet incorporates already existing information about fever, alarm symptoms, advices use of medication and specific infectious diseases that frequently occur in childhood in combination with fever such as upper respiratory tract infections, and otitis media. The difference with these existing sources of information is the fact that they until now, were not incorporated into one booklet which can be physically handed over to parents.
  Other Names: Interactive booklet
  Arms: Intervention

SUMMARY:
The CHILI cluster randomised controlled trial (RCT) will investigate whether the use of an interactive information booklet during consultations for febrile children at General Practice (GP) out-of-hours centres can reduce the number of antibiotic prescriptions, improve parental satisfaction and reduce intention to reconsult for childhood fever episodes.

DETAILED DESCRIPTION:
A GP-parent information exchange tool in the form of an interactive booklet has the potential to provide parents with information about symptoms and fever management and consistent information during GP consultations. Thereby enhancing their self-management and providing them with safety net advice when they return home.

It is hypothesized that the use of such an interactive booklet during consultations for febrile children at GP out-of-hours centres will result in a reduced number of antibiotic prescriptions, improved parental satisfaction and reduced intention to re-consult.

The development of the interactive booklet concerned a three-stage process and is based on extensive qualitative work among parents, GPs and other professionals involved in childhood fever management. The booklet incorporates already existing information about fever, alarm symptoms, advice on use of medication and specific infectious diseases that frequently occur in childhood in combination with fever such as upper respiratory tract infections, and otitis media.

We will perform a cluster-randomised controlled trial at 20 GP out-of-hours centres in the Netherlands. GP out-of-hours centres will be stratified by size, to ensure equal distribution of size between the intervention and control group. The required number of clusters and participants was based on the following assumptions: (1) ICC of 0.01, (2) alpha of 0.05, power of 0.80, (3) proportion of antibiotic prescriptions in control group of 25% and a proportion of 19% in the intervention group (6% minimal clinical relevant difference) and (4) 10% loss to follow-up and 10% efficiency loss based on unequal cluster sizes. Based on a previous cohort study, we estimated to include 1000 children per cluster (GP out-of-hours centre) within six months, resulting in a need for 20 clusters and an effective sample size of 737 patients in the intervention and control group (1474 in total).

The booklet will be used during consultations with febrile children at the GP out-of-hours centres that are randomly allocated by computer to the intervention. The child's symptoms will determine which information and advice parents receive from the GP.

Statistical analysis will be performed based on intention to treat principle by performing multilevel logistic regression analysis using IBM SPSS version 21.0 and MLwiN software. We will determine independent factors associated with antibiotic prescriptions. The same will be done for secondary outcomes.

All data will be obtained, managed and monitored according to the guidelines of Good Clinical Practice.

ELIGIBILITY:
Inclusion Criteria:

* Age between three months and twelve years
* GP decides this is a fever-related consultation

Exclusion Criteria:

* Age under 3 months or over 12 years
* GP decides this is NOT a fever-related consultation

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1262 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Antibiotic Prescription | Baseline (Initial consultation)
  Antibiotic prescriptions for febrile children in GP out-of-hours centres during the initial consultation (dichotomous scale; number of participants with an antibiotic prescription).

SECONDARY OUTCOMES:
Intention to re-consult | Asked within two weeks after initial consultation
  Intention to re-consult for similar illnesses among parents, number of parents with the intention to re-consult
Parental satisfaction with care | Asked within two weeks after initial consultation
  VAS scale 1-10
Self-reported adverse events related to the fever episode like hospital admission | Asked within two weeks after initial consultation
Antibiotic prescription rates at re-consultations | Asked within two weeks after initial consultation
  Prescription rates at re-consultations for the same illness episode (defined as a consultation for the same reason over the last two weeks)
Consultation rates | During complete study period, during 6 months of study completion
  Consultation rates of fever related consultations of children below the age of 12 years between intervention and control groups, through 6 months of study completion.
Referral to secondary care | Baseline (during initial consultation)
  Number of participants with Referral to secondary care during initial consultation

CONTACTS AND LOCATIONS:
Overall Officials: Eefje de Bont, MD, MSc, Principal Investigator — Research Institute CAPHRI, Department of Family Medicine, Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] de Bont EG, Alink M, Falkenberg FC, Dinant GJ, Cals JW. Patient information leaflets to reduce antibiotic use and reconsultation rates in general practice: a systematic review. BMJ Open. 2015 Jun 3;5(6):e007612. doi: 10.1136/bmjopen-2015-007612. PMID 26041493
- [Background] de Bont EG, Lepot JM, Hendrix DA, Loonen N, Guldemond-Hecker Y, Dinant GJ, Cals JW. Workload and management of childhood fever at general practice out-of-hours care: an observational cohort study. BMJ Open. 2015 May 19;5(5):e007365. doi: 10.1136/bmjopen-2014-007365. PMID 25991452
- [Background] de Bont EG, Peetoom KK, Moser A, Francis NA, Dinant GJ, Cals JW. Childhood fever: a qualitative study on GPs' experiences during out-of-hours care. Fam Pract. 2015 Aug;32(4):449-55. doi: 10.1093/fampra/cmv029. Epub 2015 Apr 25. PMID 25914101
- [Background] de Bont EG, Cals JW. [An individual 'traffic light system' for children with fever?]. Ned Tijdschr Geneeskd. 2014;158:A7649. Dutch. PMID 24754933
- [Background] de Bont EG, van Loo IH, Dukers-Muijrers NH, Hoebe CJ, Bruggeman CA, Dinant GJ, Cals JW. Oral and topical antibiotic prescriptions for children in general practice. Arch Dis Child. 2013 Mar;98(3):228-31. doi: 10.1136/archdischild-2012-303134. Epub 2012 Dec 25. PMID 23268371
- [Background] de Bont EG, Loonen N, Hendrix DA, Lepot JM, Dinant GJ, Cals JW. Childhood fever: a qualitative study on parents' expectations and experiences during general practice out-of-hours care consultations. BMC Fam Pract. 2015 Oct 7;16:131. doi: 10.1186/s12875-015-0348-0. PMID 26446754
- [Derived] de Bont EGPM, Dinant GJ, Elshout G, van Well G, Francis NA, Winkens B, Cals JWL. Booklet for Childhood Fever in Out-of-Hours Primary Care: A Cluster-Randomized Controlled Trial. Ann Fam Med. 2018 Jul;16(4):314-321. doi: 10.1370/afm.2265. PMID 29987079
- [Derived] de Bont EG, Dinant GJ, Elshout G, van Well G, Francis NA, Winkens B, Cals JW. An illness-focused interactive booklet to optimise management and medication for childhood fever and infections in out-of-hours primary care: study protocol for a cluster randomised trial. Trials. 2016 Nov 17;17(1):547. doi: 10.1186/s13063-016-1667-8. PMID 27855719